CLINICAL TRIAL: NCT01994759
Title: Optimal Treatment of Plantar Fasciitis: A Randomized Clinical Trial Using Physical Training, Glucocorticoid Injections or a Combination Thereof.
Brief Title: Optimal Treatment of Plantar Fasciitis: Physical Training, Glucocorticoid Injections or a Combination Thereof.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Fonden for Faglig Udvikling af Speciallægepraksis, Denmark (Unknown)
Responsible Party: Principal Investigator, Finn Elkjær Johannsen, chief physician, MD, specialist in Rheumatology, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2012-150-FJ
Record Dates: First submitted 2013-11-10; First posted 2013-11-26 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Plantar Fasciitis
Keywords: Plantar fasciitis; Treatment; Training; Glucocorticosteroid injection
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Methylprednisolone; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Training (Active Comparator): strengthening and stretching exercises.
  Interventions: Other: Training; Behavioral: Reduction in impact
- Glucocorticosteroid injection (Active Comparator): Injection of 40 mg methylprednisolone.
  Interventions: Drug: Glucocorticosteroid injection; Behavioral: Reduction in impact
- Training and Glucocorticosteroid injections (Active Comparator): A combination treatment of the two above.
  Interventions: Other: Training; Drug: Glucocorticosteroid injection; Behavioral: Reduction in impact

INTERVENTIONS:
Other: Training — Patients are instructed to carry out strengthening exercises for the fascia plantaris 3 days a week and stretching exercises every day. Four times in the first 2 months supervised training in groups is carried out with a physiotherapist supervising the exercises and instructing in progression and new exercises, and all participants are instructed to carry out a specific training program daily at home. The amount of training performed by each patient, is registered in a diary weekly
  Other Names: Heavy slow resistance exercise; Eccentric training; stretching
  Arms: Training; Training and Glucocorticosteroid injections
Drug: Glucocorticosteroid injection — Ultra sound guided injection af 1 ml og Glucocorticosteroid (methylprednisolone 40 mg) and 1 ml of lidocaine 5mg/ml from the medial side profound to the thickened part of the fascia plantaris.
  Glucocorticosteroid injections are given every month until the aponeurosis thickness is less than 4 mm as determined by ultrasonography (max 3 injections).
  Other Names: Methylprednisolone; Depo-medrol
  Arms: Glucocorticosteroid injection; Training and Glucocorticosteroid injections
Behavioral: Reduction in impact — advocate reduction in standing, walking, running, jumping. advocate shock absorbing shoes advocate prefabricated insoles advocate taping in special occasions.
  Other Names: Shock absorbtion

SUMMARY:
The purpose of this study is to determine whether reduced load to patients with plantar fasciitis (reduced standing, walking, landing) together with either controlled heavy resistance training or glucocorticosteroid injection or a combination thereof is the best treatment.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is a frequently diagnosed condition, defined as pain at the medial tubercle of the calcaneus, and 10% of the population will at some points in their life experience this condition. Accumulated loading of the plantar fascia seems to relate to development of PF, as it is commonly seen in runners and those who are overweight, and number of daily steps or simply time of standing has been shown to be a predisposing factor for PF development.

Orthosis and glucocorticoid injections are 2 widely used treatments with proven effect. However treatment of overuse injury in other tendon/aponeurosis-like structures, has over the later years been dominated by an increasing documentation of a good curative effect of heavy controlled mechanical loading (eccentric strength exercises or heavy slow concentric strength training) upon tendinopathies in Achilles or patella tendon. However, no studies have looked at the influence of physical training (e.g. strength training) on the diseased plantar aponeurosis. Also no studies have looked at the effect of a combination of giving local glucocorticoid injection and training on this or other tendon overuse entities.

We hypothesize that heavy strength training will have a positive effect upon PF, and that a combination of training and glucocorticoid injections will have an additive effect upon this disease and be even more effective than each of the treatments alone. Glucocorticoid injection acting as the standard control treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pain at the medial attachment of fascia plantaris.
* First step pain in the morning
* Symptoms for at least 3 months.
* Age 20-65 years
* Ultrasound scanning at the first visit shows thickness of the fascia above 4 mm.
* Patient can read and understand danish

Exclusion Criteria:

* known arthritis, inflammatory bowl disease, psoriasis or clinical signs of any of these
* Leg ulcerations
* Longlasting oedema of the leg and foot
* Palpatory decreased puls in the foot
* Diabetes
* Reduced sensibility in the foot
* Infections in the foot
* Daily use of pain killers
* Pregnancy or planning to become pregnant
* Earlier operations on the foot, that is judged to complicate training
* Patient assessed not to be able to participate in the training for other reasons
* Glucocorticosteroid injection to the diseased plantar fascia within the last 6 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
100 mm VAS score pain at function. Average pain during everyday living. | 6 month
Foot Function Index | 6 month
  Foot function Index is a validated score for patients with plantar fasciitis. It consists of 23 questions concerning pain, function and impact on daily life. Each question is answered on a box scale 0-10, giving a score range: 0-230.

SECONDARY OUTCOMES:
100 mm VAS score for morning pain | at entry, 3 month (after intervention), 6 month, 12 month, 24 month
Ultrasound scanning thickness measure | at entry, 3 month (after intervention), 6 month, 12 month, 24 month
  measurement of the thickness of the thickest part of the fascia by B-mode Ultrasound scanning
100 mm VAS score pain at function. Average pain during everyday living. | 3 months, 12 months, 24 months
Foot Function Index | 3 month, 12 month, 24 month
  Foot function Index is a validated score for patients with plantar fasciitis. It consists of 23 questions concerning pain, function and impact on daily life. Each question is answered on a box scale 0-10, giving a score range: 0-230.

OTHER OUTCOMES:
patient diary | week 1,2,3,4,5,6,7,8,9,10,11,12,13
  100 mm VAS score for morning pain (average in the week). 100 mm VAS score for pain at function (average in the week). Compliance to the treatment. Side effects to glucocorticosteroid injections is described.
Contrast Enhanced Ultrasound | at entry after 3-4 months and after 1 year
  For determining bloodflow of the plantar fascia we inject 2 ml SonoVue®. Ultrasound contrast agent, that amplifies the ultrasound signal. After injection we simultaneously ultrasound scan both feet for 3 minutes. The perfusion of the fascia can hereby bee calculated.
  Only patients with unilateral plantar fasciitis will bee offered this evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjær, Professor, Study Chair — University of Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Baldassin V, Gomes CR, Beraldo PS. Effectiveness of prefabricated and customized foot orthoses made from low-cost foam for noncomplicated plantar fasciitis: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Apr;90(4):701-6. doi: 10.1016/j.apmr.2008.11.002. PMID 19345789
- [Background] Crawford F, Thomson C. Interventions for treating plantar heel pain. Cochrane Database Syst Rev. 2003;(3):CD000416. doi: 10.1002/14651858.CD000416. PMID 12917892
- [Background] Uden H, Boesch E, Kumar S. Plantar fasciitis - to jab or to support? A systematic review of the current best evidence. J Multidiscip Healthc. 2011;4:155-64. doi: 10.2147/JMDH.S20053. Epub 2011 May 24. PMID 21655342
- [Background] Vohra PK, Kincaid BR, Japour CJ, Sobel E. Ultrasonographic evaluation of plantar fascia bands. A retrospective study of 211 symptomatic feet. J Am Podiatr Med Assoc. 2002 Sep;92(8):444-9. doi: 10.7547/87507315-92-8-444. PMID 12237265
- [Background] Tobin L, Simonsen L, Bulow J. Real-time contrast-enhanced ultrasound determination of microvascular blood volume in abdominal subcutaneous adipose tissue in man. Evidence for adipose tissue capillary recruitment. Clin Physiol Funct Imaging. 2010 Nov;30(6):447-52. doi: 10.1111/j.1475-097X.2010.00964.x. Epub 2010 Aug 22. PMID 20731685
- [Background] Roos E, Engstrom M, Soderberg B. Foot orthoses for the treatment of plantar fasciitis. Foot Ankle Int. 2006 Aug;27(8):606-11. doi: 10.1177/107110070602700807. PMID 16919213
- [Background] Radford JA, Landorf KB, Buchbinder R, Cook C. Effectiveness of low-Dye taping for the short-term treatment of plantar heel pain: a randomised trial. BMC Musculoskelet Disord. 2006 Aug 9;7:64. doi: 10.1186/1471-2474-7-64. PMID 16895612
- [Background] Pfeffer G, Bacchetti P, Deland J, Lewis A, Anderson R, Davis W, Alvarez R, Brodsky J, Cooper P, Frey C, Herrick R, Myerson M, Sammarco J, Janecki C, Ross S, Bowman M, Smith R. Comparison of custom and prefabricated orthoses in the initial treatment of proximal plantar fasciitis. Foot Ankle Int. 1999 Apr;20(4):214-21. doi: 10.1177/107110079902000402. PMID 10229276
- [Background] Kongsgaard M, Kovanen V, Aagaard P, Doessing S, Hansen P, Laursen AH, Kaldau NC, Kjaer M, Magnusson SP. Corticosteroid injections, eccentric decline squat training and heavy slow resistance training in patellar tendinopathy. Scand J Med Sci Sports. 2009 Dec;19(6):790-802. doi: 10.1111/j.1600-0838.2009.00949.x. Epub 2009 May 28. PMID 19793213
- [Background] Cheng JW, Tsai WC, Yu TY, Huang KY. Reproducibility of sonographic measurement of thickness and echogenicity of the plantar fascia. J Clin Ultrasound. 2012 Jan;40(1):14-9. doi: 10.1002/jcu.20903. Epub 2011 Nov 22. PMID 22109854
- [Derived] Johannsen FE, Herzog RB, Malmgaard-Clausen NM, Hoegberget-Kalisz M, Magnusson SP, Kjaer M. Corticosteroid injection is the best treatment in plantar fasciitis if combined with controlled training. Knee Surg Sports Traumatol Arthrosc. 2019 Jan;27(1):5-12. doi: 10.1007/s00167-018-5234-6. Epub 2018 Nov 15. PMID 30443664